CLINICAL TRIAL: NCT00258557
Title: Phase III Randomized, Controlled, Open-label Trial to Investigate the Antiviral Activity, Tolerability and Safety of TMC114/r in Treatment- Naive HIV-1 Infected Patients.
Brief Title: TMC114-C211: Trial of an Investigational Protease Inhibitor TMC114 With Ritonavir ("TMC114/r") in HIV-1 Infected Patients Who Have Never Been Treated With Antiretroviral Medications.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002800; TMC114-C211 (Other: Tibotec Pharmaceuticals, Ireland)
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: HIV
Keywords: HIV; Anti-Retroviral agents; HIV-1; TMC114/r; Treatment naïve patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 002 (Experimental): TMC-114/RTV two 400 mg tablets of TMC114 + one 100 mg capsule of RTV daily for max. 192 weeks
  Interventions: Drug: TMC-114/RTV
- 001 (Active Comparator): LPV/RTV 400/100 mg twice daily or 800/200 mg daily depending on the country for max. 192 weeks
  Interventions: Drug: LPV/RTV

INTERVENTIONS:
Drug: LPV/RTV — 400/100 mg twice daily or 800/200 mg daily depending on the country for max. 192 weeks
  Arms: 001
Drug: TMC-114/RTV — two 400 mg tablets of TMC114 + one 100 mg capsule of RTV daily for max. 192 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to compare the efficacy, safety and tolerability of TMC114/r versus Kaletra (a combination pill of lopinavir and ritonavir, ("lpv/rtv") in HIV-1 infected patients who have never been treated with anti-retroviral medications (referred to as "treatment-naïve" patients).

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label trial to investigate the antiviral activity, tolerability and safety of TMC114/r) versus lpv/rtv in treatment-naive HIV-1 infected patients. Six hundred sixty treatment-naïve HIV-1 infected patients will be randomized in a 1:1 ratio to either 800/100 mg of TMC114/r once daily, or a total daily dose of 800/200 mg of lpv/rtv. All patients will take TMC114/r or lpv/rtv in combination with an NRTI background of Truvada (a combination pill of tenofovir and emtricitabine, "TDF/FTC"). The trial will consist of a screening period of approximately 14 to 28 days and a 96-week treatment period, followed by a 4-week follow-up period. The anti HIV-1 therapy initiated at baseline cannot be changed until the end of the treatment period. After the end of the treatment period (maximum of 96 weeks), patients will be followed for an additional 4 weeks to follow-up on any adverse events or laboratory abnormalities until resolution. Patients who fail either virologically or due to intolerance from the TMC114/r or lpv/rtv therapy, as judged by the investigator, or who meet one of the withdrawal criteria will be withdrawn from the trial and may have the opportunity to participate in the rollover phase of the trial.

The primary efficacy parameter is virologic response defined as a confirmed viral load < 50 copies/mL at Week 48 the objective of this study is to establish non-inferiority of TMC114/r versus lpv/rtv in terms of virologic response at Week 48 using a non-inferiority margin of 12%. To test this hypothesis, a two-sided 95% confidence interval (CI) of the difference in response rate between TMC114/r and lpv/rtv will be derived: If the lower bound of the CI exceeds -12%, non-inferiority will be concluded. Patients will take oral doses for up to 96 weeks of either 800/100mg of TMC114/r 1x/day or 800/200mg of lpv/rtv once daily, each in combination with TDF/FTC. (The 400/100 mg 2x/day dose of lpv/rtv will be used where the 1x/day use of lpv/rtv is not approved).

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented HIV-1 infection
* Screening plasma HIV-1 RNA >= 5000 copies/mL
* Patients qualify for treatment initiation based on the investigator's assessments and/or according to treatment guidelines
* Patients who can comply with the protocol requirements
* General medical condition, in the investigator's opinion, does not interfere with the assessments and the completion of the trial.

Exclusion Criteria:

* Presence of any currently active AIDS defining illness or receiving treatment for primary HIV infection
* Life expectancy of less than 6 months
* Previous or current use of antiretroviral medications (ARVs) for the treatment of HIV-infection or hepatitis B infection with anti-HIV activity
* Female -patients who are pregnant or breast-feeding, or are of childbearing potential without use of effective non-hormonal birth control methods or not willing to continue practicing these birth control methods for at least 30 days after the end of the treatment period
* -patients with a grade 3 or 4 laboratory abnormality as defined by DAIDS grading, or a calculated creatinine clearance (CLCr) < 70 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Confirmed Virologic Response defined as a Viral Load < 50 copies/mL at Week 48 | 48 weeks

SECONDARY OUTCOMES:
Evaluation of safety, tolerability, and durability of efficacy over 96 weeks of treatment | 192 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (89):
- United States (24):
  - Phoenix, Arizona
  - Beverly Hills, California
  - Long Beach, California
  - Los Angeles, California
  - Sacramento, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Orlando, Florida
  - Safety Harbor, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Las Vegas, Nevada
  - Brooklyn, New York
  - Chapel Hill, North Carolina
  - Winston-Salem, North Carolina
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Houston, Texas
- Argentina (3):
  - Buenos Aires
  - Mar del Plata
  - Neuquén
- Australia (4):
  - Brisbane
  - Darlinghurst
  - Surry Hills
  - Westmead
- Vienna, Austria
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Canada (4):
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Chile (2):
  - Providencia
  - Santiago
- Costa Rica (2):
  - Costa Rica
  - San José
- Denmark (3):
  - Aalborg
  - Copenhagen Ø
  - Hvidovre
- France (5):
  - Bobigny
  - Lyon
  - Nice
  - Orléans
  - Paris
- Germany (8):
  - Berlin
  - Cologne
  - Erlangen
  - Freiburg im Breisgau
  - Hamburg
  - Mannheim
  - Munich
  - München
- Athens, Greece
- Guatemala City, Guatemala
- Sungai Buloh, Malaysia
- Mexico (4):
  - Del Tlalpan
  - Guadalajara
  - Mex Ctity
  - Mexico City
- Panama City, Panama
- San Juan, Puerto Rico
- Russia (7):
  - Kazan'
  - Krasnodar
  - Moscow
  - Saint Petersburg
  - Smolensk
  - Volgograd
  - Voronezh
- Singapore, Singapore
- South Africa (4):
  - Cape Town
  - Dundee
  - Johannesburg
  - Pretoria
- Barcelona, Spain
- Zurich, Switzerland
- Taiwan (2):
  - Taipei
  - Tiachung
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
- United Kingdom (2):
  - Brighton
  - London

REFERENCES:
- [Result] Mills AM, Nelson M, Jayaweera D, Ruxrungtham K, Cassetti I, Girard PM, Workman C, Dierynck I, Sekar V, Abeele CV, Lavreys L. Once-daily darunavir/ritonavir vs. lopinavir/ritonavir in treatment-naive, HIV-1-infected patients: 96-week analysis. AIDS. 2009 Aug 24;23(13):1679-88. doi: 10.1097/QAD.0b013e32832d7350. PMID 19487905
- [Derived] Orkin C, DeJesus E, Khanlou H, Stoehr A, Supparatpinyo K, Lathouwers E, Lefebvre E, Opsomer M, Van de Casteele T, Tomaka F. Final 192-week efficacy and safety of once-daily darunavir/ritonavir compared with lopinavir/ritonavir in HIV-1-infected treatment-naive patients in the ARTEMIS trial. HIV Med. 2013 Jan;14(1):49-59. doi: 10.1111/j.1468-1293.2012.01060.x. Epub 2012 Oct 23. PMID 23088336
- See also: Phase III randomized, controlled, open-label trial to investigate the antiviral activity, tolerability and safety of TMC114/r in treatment- naive HIV-1 infected patients. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=988&filename=CR002800_CSR1.pdf
- See also: Phase III randomized, controlled, open-label trial to investigate the antiviral activity, tolerability and safety of TMC114/r in treatment- naive HIV-1 infected patients. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=988&filename=CR002800_CSR2.pdf